CLINICAL TRIAL: NCT04251052
Title: A Non-Randomized Prospective Clinical Trial Comparing the Non-Inferiority of Salpingectomy to Salpingo-oophorectomy to Reduce the Risk of Ovarian Cancer Among BRCA1 Carriers [SOROCk]
Brief Title: A Study to Compare Two Surgical Procedures in Individuals With BRCA1 Mutations to Assess Reduced Risk of Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NRG-CC008; NCI-2019-07791 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC008 (Other: NRG Oncology); NRG-CC008 (Other: DCP); NRG-CC008 (Other: CTEP); UG1CA189867 (NIH)
Record Dates: First submitted 2020-01-14; First posted 2020-01-31 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Ovariectomy; Specimen Handling; Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: This is a non-randomized prospective trial to determine if bilateral salpingectomy (BLS) is non-inferior to bilateral salpingo-oophorectomy (BSO) in terms ovarian, primary peritoneal, and fallopian tube cancer risk among gBRCA1m carriers between 35 and 50 years old. Individuals choose the treatment they want to receive in collaboration with their physician(s).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (bilateral salpingectomy) (Experimental): Patients undergo bilateral salpingectomy. Patients may then undergo oophorectomy after initial surgery. Patients also undergo a pelvic or transvaginal ultrasound or pelvic MRI during screening and blood sample collection throughout the trial.
  Interventions: Procedure: Bilateral Salpingectomy; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Transvaginal Ultrasound; Procedure: Ultrasound Imaging
- Group II (bilateral salpingo-oophorectomy) (Active Comparator): Patients undergo bilateral salpingo-oophorectomy. Patients also undergo a pelvic or transvaginal ultrasound or pelvic MRI during screening and blood sample collection throughout the trial.
  Interventions: Procedure: Bilateral Salpingectomy with Oophorectomy; Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Transvaginal Ultrasound; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Bilateral Salpingectomy — Undergo bilateral salpingectomy
  Arms: Group I (bilateral salpingectomy)
Procedure: Bilateral Salpingectomy with Oophorectomy — Undergo bilateral salpingo-oophorectomy
  Other Names: bilateral salpingo-oophorectomy
  Arms: Group II (bilateral salpingo-oophorectomy)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Magnetic Resonance Imaging — Undergo pelvic MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Transvaginal Ultrasound — Undergo transvaginal ultrasound
  Other Names: transvaginal sonography; TVS; TVU
Procedure: Ultrasound Imaging — Undergo pelvic ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This clinical trial evaluates how well two surgical procedures (bilateral salpingectomy and bilateral salpingo-oophorectomy) work in reducing the risk of ovarian cancer for individuals with BRCA1 mutations. Bilateral salpingectomy involves the surgical removal of fallopian tubes, and bilateral salpingo-oophorectomy involves the surgical removal of both the fallopian tubes and ovaries. This study may help doctors determine if the two surgical procedures are nearly the same for ovarian cancer risk reduction for women with BRCA1 mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the non-inferiority of bilateral salpingectomy (BLS) with delayed oophorectomy to bilateral salpingo-oophorectomy (BSO) to reduce the risk of ovarian cancer among individuals with deleterious BRCA1 germline mutations.

SECONDARY OBJECTIVES:

I. To prospectively assess estrogen deprivation symptoms in pre-menopausal BLS patients as measured by the Functional Assessment of Cancer Therapy - Endocrine Symptom (FACT-ES) subscale compared to pre-menopausal patients in the BSO arm.

II. To determine if health-related quality of life (QOL) (FACT) is negatively impacted by menopausal symptoms (menopausal symptom checklist-Menopausal Symptom Checklist [MSCL]) and sexual dysfunction (Female Sexual Function Index [FSFI]) in pre-menopausal patients who have undergone BLS, in comparison to normative data (MSCL/FACT-ES) and data from pre-menopausal BSO patients.

III. To determine if health-related QOL (FACT) is negatively impacted by cancer distress (Impact of Event Scale [IES]) in individuals who have undergone BLS, in comparison to BSO patients.

IV. To assess medical decision making, as measured by the Shared Decision Making Questionnaire (SDM-Q-9) and Decision Regret Scale (DRS), and determine factors associated with the risk of reducing surgical treatment choice.

V. To assess adverse events, graded using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

EXPLORATORY OBJECTIVES:

I. Sexual dysfunction, as measured by selected Patient-Reported Outcomes Measurement Information System (PROMIS) screener and external sexual function items (pre-menopausal patients).

II. To estimate the cost-effectiveness of BLS compared to BSO for ovarian cancer risk reduction.

III. To assess medical decision making, as measured by the Risk-Reducing Medical Decision Making (RR-MDM) survey, a targeted set of questions on risk reducing surgical treatment choice.

TRANSLATIONAL RESEARCH OBJECTIVE:

I. To bank tissue and blood biospecimens for future research.

OUTLINE: Patients choose between 1 of 2 groups.

GROUP I: Patients undergo bilateral salpingectomy. Patients may then undergo oophorectomy after initial surgery.

GROUP II: Patients undergo bilateral salpingo-oophorectomy.

Patients in both groups also undergo a pelvic or transvaginal ultrasound or pelvic magnetic resonance imaging (MRI) during screening and blood sample collection throughout the trial.

After completion of study, patients are followed up at 10-60 days, 6, 12, and 24 months, and then annually for up to 20 years.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 35-50 years of age, inclusive
* Patients who will undergo risk-reducing salpingo-oophorectomy (RRSO) (for the BSO arm) and patients who have declined or elected to defer BSO after proper counselling to clearly explain the standard of care for BRCA1 mutation carriers and are undergoing salpingectomy (for the BLS arm with delayed oophorectomy arm). Concurrently planned hysterectomy with either arm is permitted
* At least one intact ovary and fallopian tube is in situ at the time of counseling, consent, and registration. Prior hysterectomy is allowed provided it did not include bilateral salpingectomy. Prior tubal ligation is allowed if one ovary and fallopian tube (with fimbria not removed) are present
* Positive Clinical Laboratory Improvement Act (CLIA)-approved test results for pathogenic or likely pathogenic germline BRCA1 mutation in the patient. Documentation of the result is required
* Patients may be premenopausal or menopausal
* Pelvic ultrasound (transvaginal imaging preferred, but transabdominal imaging is acceptable) or pelvic MRI and CA-125 within 180 days of registration
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Individuals who are currently pregnant or plan to become pregnant in the future through assisted reproductive technologies and who have received proper counseling are eligible. Individuals who are currently pregnant and plan bilateral salpingectomy at the time of a planned cesarean section are eligible. Patients must understand that they will not be able to become pregnant naturally in the future

Exclusion Criteria:

* Individuals with a history of any prior cancer who have received cytotoxic chemotherapy within the past 30 days or radiotherapy to abdomen or pelvis at any prior time. Endocrine therapy or maintenance ERBB2/HER2 targeted therapy is allowed. Maintenance immune checkpoint inhibitor therapy is allowed. Maintenance therapy with PARP in inhibitor is allowed.
* Prior history of ovarian cancer, including low malignant potential neoplasms (LMP), primary peritoneal carcinoma, or fallopian tube carcinoma
* Patients medically unfit for the planned surgical procedure
* Patients with abnormal screening tests (pelvic ultrasound, pelvic MRI, CA-125) suspicious for occult or gross pelvic malignancy within the past 180 days

  * An abnormal pelvic ultrasound (or pelvic MRI) is defined as morphologic or structural variations suspicious for ovarian malignancy. Complex cystic lesions felt to represent a benign lesion are not exclusionary. Simple cysts of any size are not exclusionary
  * An abnormal CA-125 is defined as a level > 50U/ml in premenopausal individuals if they are not current users of oral contraceptives; an abnormal CA-125 is defined as a level > 40U/ml for premenopausal individuals who are current users of oral contraceptives (Skates 2011). An abnormal CA-125 is defined as a level > 35 U/ml in postmenopausal individuals

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1956 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2047-06-30 (Estimated); Study Completion 2047-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to development of incident high-grade serous carcinomas (HGSC), specifically ovarian, primary peritoneal, or fallopian tube cancers | Up to 20 years
  Will be assessed using a stratified log rank test, stratifying for age. The effects of other covariates, such as familial history of gynecologic cancer, time to crossover for bilateral salpingectomy (BLS) patients, and age at study entry, will be adjusted for in Cox proportional hazard models. Patients who crossover will be analyzed according to the initial surgery received at study enrollment as this will reflect actual practice.

SECONDARY OUTCOMES:
Health-related quality of life (QOL) | Up to 24 months post-surgery
  Will be measured by the Functional Assessment of Cancer Therapy - Endocrine Symptom (FACT-ES). The FACT total score (calculated from the physical, functional, social and emotional well-being subscales) and ES subscale will be assessed. Scores range from 0 to 76. Higher scores indicate better QOL for the FACT-ES and better functioning for the Female Sexual Function Index (FSFI) total score.
Cancer distress | Up to 24 months post-surgery
  Will be measured by the Impact of Events Scale (IES). The total score can range from 0 to 88, with higher scores indicating a greater impact of the event.
Medical decision making | Up to 24 months post-surgery
  Will be measured by the Shared Decision Making Questionnaire (SDM-Q-9) and, Decisional Regret Scale. The SDM-Q-9 total score and Decisional Regret Scale total score at each time point of collection will be compared between arms using a t-test with a significance level of 0.05. A linear model will be used to assess the association of the SDM-Q-9 total score with treatment arm and patient characteristics such as age and race. A similar model will be used to assess the association of the Decisional Regret Scale total score with treatment arm and patient characteristics such as age, race, crossover from BLS arm, and hysterectomy status. Minimum score of 0 and a maximum score of 45. A higher score indicates a greater level of perceived shared decision-making in a consultation.
Incidence of adverse events | Up to 20 years
  Will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Counts and frequencies will be provided for the worst grade adverse event (AE) experienced by the patient by treatment arm. The distribution of AE grade in the BLS arm will be compared to the bilateral salpingo-oophorectomy arm using a chi-square test, or Fisher's exact test if cell frequencies are < 5, at the one-sided 0.05 significance level.
Estrogen deprivation symptoms (pre-menopaused patients only) | Up to 24 months post-surgery
  Will be measured by the FACT-ES. The FACT total score (calculated from the physical, functional, social and emotional well-being subscales) and ES subscale will be assessed. Scores range from 0 to 76. Higher scores indicate better QOL for the FACT-ES and better functioning for the FSFI total score. Models will also include hormonal therapy as a covariate.
Sexual dysfunction (pre-menopausal patients only) | Up to 24 months post-surgery
  Will be measured by the FSFI. Scores range from 0 to 36. Higher scores indicate better functioning for the FSFI total score.
Menopausal symptoms (pre-menopausal patients only) | Up to 24 months post-surgery
  Will be measured by the Menopausal Symptom Checklist (MSCL). Models will also include hormonal therapy as a covariate. The MSCL total score and individual items will be compared between groups using the t-test and Wilcoxon test, respectively. The change from baseline in total score will be compared between groups at each follow-up time point. The change form baseline in the 3 items not included in the subscale scores will be compared between groups using the Wilcoxon test at each follow-up time point.

OTHER OUTCOMES:
Cost effectiveness | Up to 24 months post-surgery
  Will be measured by European Quality of Life Five Dimension Five Level Scale Questionnaire. A Markov model will be used to model cost. Scores range from 0 to 100 with higher score indicating better overall health.
Sexual dysfunction (pre-menopausal patients only) | Up to 24 months-post surgery
  Will be measured by selected Patient-Reported Outcomes Measurement Information System (PROMIS) screener and external sexual function items. Each item will be analyzed separately and compared between treatment arms using a chi-square test. Scores range from 0 to 100 with higher score indicating more of the concept being measured.
Health related (HR)-QOL | Up to 24 months post-surgery
  Will examine the correlation between HR-QOL, as measured by the FACT, with menopausal symptoms, as measured by the MSCL, sexual dysfunction, as measured by FSFI, and PROMIS screener and external sexual function items and cancer distress as measured by the IES. Pearson correlation coefficients will be used for correlating the FACT total score with the FSFI overall score and Impact of Events Scale total distress score. Spearman correlation coefficients will be used to assess the correlation between FACT total score and the Menopausal Symptom Checklist symptoms, FSFI, and PROMIS items.
Risk-reducing medical decision making validation and assessment | Up to 24 months post-surgery
  Measured by population-specific items examining the factors associated with the risk reducing surgical treatment choice. Will by assessed using the Risk-Reducing Medical Decision Making survey.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn P Pennington, Principal Investigator — NRG Oncology
Locations (542):
- United States (533):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Keck Medicine of USC Buena Park, Buena Park, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - City of Hope Seacliff, Huntington Beach, California
  - Keck Medicine of USC Huntington Beach, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Providence Queen of The Valley, Napa, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Huntington Memorial Hospital, Pasadena, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Florida Cancer Specialists - Bradenton Cancer Center, Bradenton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - Florida Cancer Specialists-Englewood, Englewood, Florida
  - GenesisCare USA - FGO, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Sarasota Memorial Hospital-Venice, Nokomis, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Intercoastal Medical Group - Cattleridge II, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - First Physicians Group - Silverstein Institute at Floyd Street, Sarasota, Florida
  - First Physicians Group - Urology Robotic and Minimally Invasive Surgery, Sarasota, Florida
  - First Physicians Group-Sarasota, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Sarasota Memorial Health Care Center at University Parkway, Sarasota, Florida
  - Saint Anthony's Hospital Cancer Care Center, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Florida Cancer Specialists - Venice Island, Venice, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Carle BroMenn Outpatient Center, Bloomington, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Rush MD Anderson Cancer Center at Rush Oak Park, Oak Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MEJ, Council Bluffs, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Baptist Health Corbin, Corbin, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Baptist Health Richmond, Richmond, Kentucky
  - West Jefferson Medical Center, Marrero, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Willis-Knighton Medical and Cancer Center, Shreveport, Louisiana
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - South Shore University Hospital, Bay Shore, New York
  - Island Gynecologic Oncology, Brightwaters, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Northwell Health Physician Partners at Flushing, Flushing, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Huntington Hospital, Huntington, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Northwell Health Physician Partners, New Hyde Park, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Northwell Physician Partners at Rego Park, Rego Park, New York
  - Queens Cancer Center, Rego Park, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Mission Hospital, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - OhioHealth O'Bleness Hospital, Athens, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - OhioHealth Pickerington Methodist Hospital, Pickerington, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center at Franklin, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - Women's Cancer Center of Seattle, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- South Korea (7):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - Samsung Changwon Hospital, Seoul, Gyeongsangnam-do
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Yonsei University Health System-Severance Hospital, Seoul

REFERENCES:
- [Derived] Pennington KP, Pugh SL, Huh W, Walker JL, Jewell E, Havrilesky LJ, Carter J, Muller CY, Drapkin R, Lankes HA, Castellano T, Zamorano AS, Blank SV, Kachnic LA. Optimization of Timing for Risk-Reducing Salpingectomy and Oophorectomy. Obstet Gynecol. 2025 Jan 1;145(1):21-30. doi: 10.1097/AOG.0000000000005781. Epub 2024 Nov 7. PMID 39509704